CLINICAL TRIAL: NCT03516825
Title: Musical Neglect Training for Unilateral Visual Neglect in Right Hemispheric Stroke Patients
Brief Title: Musical Neglect Training for Patients With Visual Neglect
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Colorado State University (Other)
Responsible Party: Principal Investigator, Michael H. Thaut, Professor, University of Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-5432H
Record Dates: First submitted 2018-04-19; First posted 2018-05-04 (Actual); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Hemispatial Neglect
Keywords: Musical Neglect Training; Neurologic Music Therapy; unilateral visual neglect; hemispatial neglect; stroke; spatial perception and attention; music therapy
MeSH Terms: conditions — Perceptual Disorders; Stroke; Orientation, Spatial

STUDY DESIGN:
Intervention Model Description: The same intervention has been used for all participants (two) for this study.
Masking Description: All participants were given no information about this intervention. Participants only followed the direction by student music therapist.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Musical Neglect Training (MNT) (Experimental): A single-subject design was used. All participants took Musical Neglect Training.
  Interventions: Other: Musical Neglect Training

INTERVENTIONS:
Other: Musical Neglect Training — MNT uses musical exercises which are structured in pitch, time and tempo, and musical equipment (tone bars, keyboards, drums) configures to focus attention to the neglect visual field.
  Other Names: Neurologic Music Therapy

SUMMARY:
Music Neglect Training has been developed for patients with hemispatial neglect to improve their attention on the left side. The purpose of this study was to examine the immediate and carry-over effect of Musical Neglect Training on unilateral visual neglect. Standardized assessments (Albert's test and Line Bisection Test) were used to measure a range of visual field. A total of 6 musical exercises with tone bars which are aligned horizontally helped to improve attention and perception of the visual field on the left side.

DETAILED DESCRIPTION:
Unilateral visual neglect from right hemisphere stroke is a condition that reduces a person's ability to attend to and process stimuli in one half, mostly left side, of their environment. This perceptual processing deficit can negatively affect individuals' daily living which in turn reduces functional independence. Music has been used as a therapeutic tool in a variety of settings to promote cognitive functions. In particular, music has been used to improve attention in the left sides for patients with visual neglect. Musical Neglect Training (MNT) has been developed for patients with visual neglect to improve attention in the left side.

The purpose of this study was to examine the immediate and longer-lasting effect of Musical Neglect Training (MNT) on unilateral visual neglect. A single-subject design was used, as participants served as their own control. Two individuals participated in this study. Participants underwent six individual MNT sessions. MNT uses musical exercises which are structured in pitch, time and tempo, and musical equipment (tone bars, keyboards, drums) configures to focus attention to the neglect visual field. Two standardized assessments (Albert's and Line Bisection Test) were used. The assessments were administered immediately before and after each of the 6 MNT sessions to assess the immediate effect of MNT. Moreover, follow-up testing was done one week after their 6th session to examine the longer-lasting effects of MNT. Paired t-test was used to examine the immediate effect, and both participants showed significant improvement with Albert's Test in immediate effect.

ELIGIBILITY:
Inclusion Criteria:

* patients with visual neglect after stroke
* right-handed
* medically stable
* no previous music therapy experiences
* no hearing impairments
* no cognitive deficits

Exclusion Criteria:

* hemianopia
* previous music therapy treatment experiences

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-01-27 (Actual); Primary Completion 2016-01-28 (Actual); Study Completion 2016-01-28 (Actual)

PRIMARY OUTCOMES:
Changes of Albert's Test between before and after the sessions | Albert's test was given to participants before and after of all 6 sessions. The outcome measure was assessed two days a week for three weeks. Also, follow-up testing was done one week after their 6th session to examine the longer-lasting effects of MNT.
  The Albert's Test was scored as the number of uncrossed lines on the sheet. The test paper consisted of 18 lines on each side, and 4 lines in the center. Since the un-crossed lines have been calculated, less score indicates positive outcomes.
Changes of Line Bisection Test between before and after the sessions | Line Bisection was given to participants before and after of all 6 sessions. The outcome measure was assessed two days a week for three weeks. Also, follow-up testing was done one week after their 6th session to examine the longer-lasting effects of MNT.
  The Line Bisection Test was calculated as percentage of the deviation from the true center of the line. A different length of 17 lines were aligned horizontally on the test paper. Since the deviation from the true central point has been measured, less score indicates positive outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Thaut, PhD, Principal Investigator — University of Toronto

IPD SHARING:
Plan to Share IPD: No
IPD will not be made available to external researchers.